CLINICAL TRIAL: NCT03570853
Title: Stress Management and Resiliency Training for Physicians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Director of Research, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018P000836
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Burnout, Professional; Stress
Keywords: Resiliency
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive the 8-week SMART-3RP intervention within a few weeks of enrolling in the study.
  Interventions: Behavioral: SMART-3RP
- No Intervention (No Intervention): Participants will not receive the SMART-3RP program and will only complete study questionnaires..

INTERVENTIONS:
Behavioral: SMART-3RP — This is an 8-week, multimodal resiliency program that targets stress with 4 main components: mind-body skills (participants learn a variety of meditation techniques, mini relaxations, walking meditation, and yoga), traditional stress management techniques, healthy lifestyle behaviors (sleep, exercise, nutrition, and social support), and cognitive reappraisal and adaptive coping skills (borrowed from cognitive behavioral therapy, acceptance and commitment therapy, and positive psychology). The program consists of 8, 1.5 hour sessions.
  Other Names: Stress Management and Resiliency Training Relaxation Response Resiliency Program; Stress Management and Resiliency Training Program (SMART Program)
  Arms: Intervention

SUMMARY:
This study is to evaluate the effects of the SMART-3RP (Stress Management and Resiliency Training Relaxation Response Resiliency Program) on physician and academic faculty well-being, perceived stress, burnout, compassion, and job satisfaction.

DETAILED DESCRIPTION:
Burnout is a serious problem in healthcare, resulting in absenteeism, decreased job satisfaction, decreased empathy, anxiety, depression, increased medical errors and decreased patient satisfaction. A growing number of studies have demonstrated that programs incorporating mind-body practices increase resilience in healthcare providers and can reduce burnout and perceived stress while increasing empathy. The Benson-Henry Institute for Mind Body Medicine (BHI) has developed a clinical program for patients known as the Stress Management and Resiliency Training Relaxation Response Resiliency Program (SMART-3RP or SMART Program for short). This study is to evaluate the effect of the SMART-3RP on physician and academic faculty well-being, perceived stress, burnout, compassion, and job satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Physicians and academic faculty of Brigham and Women's Hospital and Newton-Wellesley Hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in perceived stress: pre-program vs. post-program | Approximately 2 months
  Change in score on the perceived stress scale - 10 item instrument (PSS-10) from baseline to completion of the group.

CONTACTS AND LOCATIONS:
Overall Officials: John Denninger, MD, PhD, Principal Investigator — Benson-Henry Institute for Mind Body Medicine
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: No